CLINICAL TRIAL: NCT00266903
Title: Treatment of Eisenmenger's Syndrome in Adults With Congenital Heart Disease With Pulmonary Arterial Vasodilators
Brief Title: Eisenmenger's Syndrome in Adults With CHD
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 05-118
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Disorders
Keywords: adult; congenital heart disease; Eisenmenger's Syndrome; Bosentan; Sitaxsetan; Sildenafil
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities; Heart Defects, Congenital; Eisenmenger Complex

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Review the outcome of treatment with endothelin receptor antagonists (bosentan or sitaxsetan) alone or in combination with Sildenafil (a PDE-5 inhibitor) in adult patients with pulmonary hypertension due to congenital heart disease.

DETAILED DESCRIPTION:
The primary objective of this study is to examine medical records of patients with Eisenmenger's Syndrome in order to determine the effect of endothelin receptor antagonists, alone or in combination, with Sildenafil, on symptoms of pulmonary hypertension. This review will be conducted on Standard of Care procedures such as New York Heart Association (NYHA) classification, six-minute walk exercise capacity, pulmonary pressures and oxygens saturations. Pulmonary pressures determined by echo or cardiac catheterization will be analyzed where available. We hypothesize that patients with congenital heart defects who develop ES will have an improved six-minute walk distance, improved pulmonary arterial pressures and improved oxygenation after treatment with endothelin receptor antagonists and other pulmonary vasodilators.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart disease (unoperated, palliated or repaired) Eisenmenger's syndrome Age 18 to 80

Exclusion Criteria:

* Those who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Congenital heart disease (unoperated, palliated or repaired) Eisenmenger's syndrome Age 18 to 80
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 1996-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Review the outcome of treatment with endothelin receptor antagonists (bosentan or sitaxsetan) alone or in combination with Sildenafil (a PDE-5 inhibitor) in adult patients with pulmonary hypertension due to congenital heart disease | 12 years
  Our study demonstrates that endothelin receptor blockers can be used to improve exercise tolerance, oxygenation, and functional status in adults with Eisenmenger syndrome without adverse effects. The role of newer treatment modalities such as prostacyclins, PDE inhibitors, and nitric oxide remain promising and their role needs to be investigated to help improve quality of life and life expectancy in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M. Book, MD, Principal Investigator — Emory University SOM
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States